CLINICAL TRIAL: NCT01816919
Title: Characterization of Head and Neck Malignant Tumors Using an Electronic Nose
Acronym: HNeNose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-09-0075-CTIL
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eNose breath samples (Experimental)
  Interventions: Other: collecting breath samples

INTERVENTIONS:
Other: collecting breath samples

SUMMARY:
Head and neck tumors are common in the general population especially in high risk groups of smokers and alcohol abusers, as well as after exposure to various environmental factors. Diagnosis is based on identification of patients gross disease after a physical examination and various imaging methods, and characterization of tissue mainly by fine-needle puncture (FNA) and biopsy. Determining the stage of disease is based on physical examination, imaging and tissue samples.

Using the electronic nose technology we hope to identify microscopic disease when it is suspected or in populations in risk, thus diagnose patients in the initial stages of the disease. Obviously, early diagnosis and treatment decisions will hopefully improve the prognosis.

Finding a positive correlation between the stages, levels and various tumor volume and respiratory specimens findings will classify patients more accurately and contribute to further characterization of the disease in a more accurate, rapid and non-invasive fashion.

DETAILED DESCRIPTION:
Approximately 60,000 new cases of head and neck cancer are diagnosed in the U.S. each year, accounting for about 5% of cancer cases diagnosed in North America and approximately 1-2% of cancer deaths.

Smoking and alcohol are the main risk factors for head and neck tumors and are recognized in 75% of cases. In contrast, consumption of fruits and vegetables was found to be a protective factor. The symptoms are varied and can include sore throat and / or neck, difficulty or pain in swallowing, difficulty in breathing and hoarseness, facial movement disorder and other.

Multidisciplinary decision making and treatment is important for these patients due to the complexity of treatment and short-and long-term complications resulting from chemotherapy, radiotherapy and surgical intervention.

About a third of patients are diagnosed with disease at stage 1 or 2. These patients are treated by surgery or radiation. Five years survival for patients diagnosed with stage I is around 90% and 70% for patients diagnosed with stage 2. Despite surgical and radiation treatment when patients present with locally advanced disease, only 30% -50% of them survive after five years. Therefore, many studies have been conducted in an attempt to improve prognosis. Improved results are seen in combination therapy with chemotherapy and radiation treatment.

Patient survival depends on the stage of the disease, hence the importance of early detection. Research Laboratory of Dr. Hossam Haick developed a device that simulates the human nose. The device reveals patterns of volatile organic compounds emitted by breathing cancer cells. This is why it is referred to as "electronic nose". It includes an array of tiny nanometer sized sensors connected to an electronic computation unit. Because of their small size and electrical properties, the sensors are able to "smell" the changes in the composition of the materials that characterize cancer. Discovery of bio - cancer markers using breath samples offers several advantages: a) The breath samples are not invasive; b) air exhaled contains mixtures less complex than those found in blood or urine, and c) breath tests allow direct monitoring in real-time.

In this study we want to test the reliability of the developed device in real clinical conditions. Another goal of these experiments is to characterize the differences between respiratory specimens for various disease stages and to examine whether there is a relationship between the results of the samples to tumor volume (calculated using diagnostic CT scans). Due to its simplicity, positive results will allow us to consider using the device as a screening device for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and neck tumors
2. A patient can understand, read and sign the informed consent form, signing a consent form
3. Age over 18

Exclusion Criteria:

1. Known or second primary head and neck cancer
2. Surgery to head and neck index tumor except for tumor biopsy
3. Unsteady comorbidity
4. Pregnancy
5. breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Characterization of biochemical markers in breath samples of patients with head and neck cancer by using artificial olfactory system (electronic nose). | one year